CLINICAL TRIAL: NCT05961241
Title: Pelvic Floor Muscle Function Among Running Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, PHD, senior lecturer, University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 170/22
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Urinary Stress Incontinence
Keywords: Urinary incontinence; pelvic diaphragm; women's health
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence | interventions — Running

STUDY DESIGN:
Intervention Model Description: Two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- running group (Active Comparator): women who run on a regular basis
  Interventions: Other: runnin training program
- control (Experimental): women who do not run
  Interventions: Other: runnin training program

INTERVENTIONS:
Other: runnin training program — gradual training program
  Other Names: running

SUMMARY:
This study will examine pelvic floor muscles function amongst women who run on a regular basis compared to controls. Women who do not run, will begin running protocol, and second evaluation will be performed following 2 months of training. Urinary incontinence will also be assessed.

DETAILED DESCRIPTION:
The study will include women who have been running on a regular basis over two years, at least 3 times a week for half an hour (research group) and women who do not run at all (control group). The participants will answer a personal information questionnaire (including birth and exercise background), and the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF). Outcome measures will include an evaluation of the PFM function using Vaginal palpation and abdominal ultrasound examination.

Women who do not run at all, will begin running training protocol, and second evaluation will be performed following 2 months of training.

ELIGIBILITY:
Inclusion Criteria:

* at least six months after giving birth or who have not given birth at all, The running group will recruit healthy women who run at least 3 times a week, 30 minutes, for two consecutive years.

The control group will recruit healthy women who do not physical active on a daily basis

Exclusion Criteria:

* pregnancy
* grade 3 or higher of pelvic organ prolapse.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study examines pelvic floor function among women
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
direction of urinary bladder displacement during contraction | baseline
  upward or downward displacement of urinary bladder will be measured via diagnostic ultrasound
urinary bladder displacement in millimeters | baseline
  bladder displacement will be measured via diagnostic ultrasound using the on screen caliper tool
pelvic floor muscles endurance of contraction in seconds | baseline
  time of muscle contraction will be measured during the last contraction
urinary incontinence | baseline
  International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF).

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, Prof., Principal Investigator — University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel